CLINICAL TRIAL: NCT02809300
Title: Prevalence of Antiphospholipid Antibodies in Ankylosing Spondylitis: A Study of 80 Patients
Brief Title: Ankylosing Spondylitis and Antiphospholipid Antibodies
Acronym: ASAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA15075
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Ankylosing Spondylarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Blood Specimen Collection

ARMS (1):
- ankylosing spondylarthritis (Experimental)
  Interventions: Biological: blood collection

INTERVENTIONS:
Biological: blood collection

SUMMARY:
The main objective is to evaluate the prevalence of anti-phospholipid antibodies (APLA) in patients with ankylosing spondylitis (AS).

The secondary objectives are: (1) To determine whether the presence of these antibodies is symptomatic (thrombosis or not); (2) Identify a possible relationship between the presence of APLA and a particular form of SA (axial or peripheral); (3) To determine whether the presence of APLA is more frequent in patients receiving anti-tumor necrosis factor (TNF) alpha therapy.

DETAILED DESCRIPTION:
Methods:

Experimental design: longitudinal study prospective in a single center.

The Ankylosing Spondylitis Assesment Study (ASAS) criteria are: (1) age <45 years, back pain ≥ 3 months, sacroiliitis on imaging and ≥ 1 associated minor criterion, or (2) HLA B27 positive and ≥ 2 minor criteria.

Minor criteria are: inflammatory back pain, arthritis, enthesitis, uveitis, Dactylitis, psoriasis, Crohn's disease, good clinical response to NSAIDs, family history of Human Leukocyte Antigen HLA B27 and inflammatory syndrome.

Plan Investigation:

Patients in the study will be seen first in consultation to gather the necessary information: history taking (including venous and arterial embolic events and obstetric history), the usual treatment, ASAS criteria of therapeutic AS, current and previous, comprehensive physical examination.

APLA will be measured at baseline and at least 3 months if initially positive.

OUTCOME:

The primary endpoint is the presence or absence of APLA: anti-cardiolipin antibodies (CLA) immunoglobulin M (IgM) or immunoglobulin G (IgG), circulating anticoagulant lupus (CCA), anti-beta2 glycoprotéine1 antibodies (β2GP1A) IgM or IgG.

The secondary endpoints are:

* The presence of thrombosis (past or present) or obstetrical accident (anterior)
* Relationship between the presence of APLA and a particular form of AS (axial or peripheral)
* Relationship between the presence of APLA and anti-TNF alpha therapy

Calendar:

The expected study duration is 16 months.

Statistical Analysis Plan A descriptive analysis will be performed. The variables are described by their number and percentage; quantitative variables are described by their mean and standard deviation. A calculation of the prevalence of APLA will be made. Univariate analysis will be performed for the secondary objectives by the Chi 2 test or Fisher exact test according to the application conditions.

ELIGIBILITY:
Inclusion criteria patients :

* older than 18 years
* with SA according to ASAS criteria
* followed in the Internal Medicine Department of the REIMS University Hospital
* who have given their consent
* affiliated to social security insurance

Exclusion criteria patients :

* minor patients
* patients with autoimmune disease (except the inflammatory bowel disease)
* cancer
* coagulation disorders
* anticoagulant treatment (anticoagulation out for events history thrombus embolism)
* pregnant women
* patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
presence or absence of APLA | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France